CLINICAL TRIAL: NCT04816903
Title: Gyni™ System Pilot Study With Leumit Health Services - Prospective Study
Brief Title: Gyni™ Study With Leumit Health Services
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GynTools Ltd. (Industry)
Collaborators: Leumit Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CL00000-16
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Vaginitis
Keywords: gynecology; IVD
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Intervention Model Description: Group-A Blinded Group-B Unblinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Symptomatic vaginitis patients (Experimental): All participants will be enrolled according to their complaints, All will be tested by the Gyni system, Only in the second group the physician will be unblinded to the Gyni results.
  Interventions: Diagnostic Test: Gyni

INTERVENTIONS:
Diagnostic Test: Gyni — Vaginal discharge collection

SUMMARY:
About one third of the women referring to gynecological clinics present with vulvovaginal inflammation symptoms (vaginitis) possibly caused by seven different conditions or mixed infections. The Gyni™ system is intended to provide physicians with the means to obtain an accurate, fast and inexpensive diagnosis which is unavailable today.

Gyni™ is comprised of a compact tabletop scanner, a disposable sample collector and a cloud based algorithm that provides a suggested diagnosis within 5 minutes.

The trial is a prospective evaluation of the cost-effectiveness of using Gyni™ by comparing its usage outcomes in a practice setting to the outcomes obtained using the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Female ≥18 years old
* Able to read, understand and sign an informed consent form
* At least one of the following: abnormal vaginal discharge, odor, vulvovaginal itch, burning, irritation, dyspareunia, vaginal dryness or pain.

Exclusion Criteria:

* Patients under the age of 18 years
* Patient is unfit to provide an informed consent
* Patient with vaginal bleeding, including menstruation within past 24 hours21
* Patient who used intra vaginal preparations within 72 hours prior to study enrollment (antimicrobials, spermicides, lubricants, diaphragm)22
* Uninterpretable sample (e.g. patients who used vaginal creams or lubricants before the visit or insufficient sampling material)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 600 (Estimated)
Dates: Start 2021-03-07 (Actual); Primary Completion 2022-03-07 (Estimated); Study Completion 2022-03-07 (Estimated)

PRIMARY OUTCOMES:
Comparison parameter | 12 months
  Number of visits (from initial visit until the cause of vaginitis is detected)
Comparison parameter | 12 months
  Total cost of medication
Comparison parameter | 12 months
  Total Cost of lab tests

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Netanya Women's health center, Leumit Health services (HMO), Netanya, Central District
  - Kfar Yasif clinic, Kfar Yasif, North
  - Kiryat Bialik, Leumit health services (HMO) Women's health clinic, Kiryat Bialik, North
  - Leumit women's health, Jerusalem

IPD SHARING:
Plan to Share IPD: No